CLINICAL TRIAL: NCT03392857
Title: End Of Life in the Critically Ill patiEnt
Acronym: EOLE
Status: Completed | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Collaborators: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EOLE
Record Dates: First submitted 2017-12-18; First posted 2018-01-08 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Terminal Illness; Intensive Care Unit Syndrome
Keywords: Critical care
MeSH Terms: interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment by caregivers of the quality of the end of life in intensive care units — Quality of the end of life in intensive care units perception will be explore from the side of the caregivers, trough the CAESAR scale.

SUMMARY:
The purpose of this multicentric study is to evaluate the perception of the quality of the end of life in intensive care units seen from the side of the caregivers, trough the CAESAR scale.

DETAILED DESCRIPTION:
More than 20% of deaths occur in hospital after a stay in intensive care units; up to half of them happens as result of a treatment limitation. Ensuring end-of-life quality is important, not only because is a moral duty of all caregivers, but also to prevent negative effects in close relatives of dead patients.

In an assessment of quality of in-hospital deaths involving 3793 patients, only 35% of the deaths were judged to be of acceptable quality by the nurses.

Assessment tools have been developed recently on this topic. Most studies have focused on the perception of end-of-life quality by close relatives, particularly through the CAESAR scale in the most recent one.

The main purpose of this multicentric study is to evaluate the perception of the quality of the end-of-life in intensive care units seen from the side of the caregivers, in relation to the new French legislative framework.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of intensive care unit whose patient has recently deceased

Exclusion Criteria:

* Refusal of participation by caregivers
* Refusal of participation by family of deceased patient
* Patient in cardiac arrest at the time of ICU admission.
* Age of deceased patient was under 18 years
* Patient in brain death

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Caregivers of patients admitted in ICU and dead in ICU.
Sampling Method: Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
15 items questionnaire CAESAR | Depending of end-of-life duration, usually 6 hours.
  The CAESAR scale assesses perceptions of palliative stage of patient's pathology, of patient's comfort, of presence and care of close relatives, with a score for each item ranging from 1 (traumatic experience) to 5 (soothing). The purpose of our study is to assess the perception of end-of-life quality seen from the caregivers' side, using the CAESAR scale.

SECONDARY OUTCOMES:
Variables associated with the perception by caregivers of end-of-life quality | time needed for the enrollment of caregivers of 5 to 15 consecutive deceased patients per center (depending on the size of the center): usually 1 month
  Evaluate the variables associated with the perception by caregivers of end-of-life quality: proportion of treatment limitations, frequencies of conflicts between close relatives of dead patients and caregivers, frequencies end-of-life deep sedations, detailed description of current sedation practices, proportion of treatments, monitoring and blood tests maintained after treatment limitation during end-of-life .
Analogic visual scale (0 to 10) | Depending of end-of-life duration, usually 6 hours.
  Analogic visual scale on end-of-life quality seen from the caregiver's side

CONTACTS AND LOCATIONS:
Overall Officials: Florence Boissier, MD, Study Director — French Intensive Care Society
Locations (111):
- France (111):
  - Hôpital Saint-Esprit, Agen
  - Centre Hospitalier Alès en Cévennes, Alès
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - Hopital Privé d'Antony, Antony
  - CH d'Argenteuil, Argenteuil
  - Hopital Mercy, Ars-Laquenexy
  - Centre Hospitalier René Dauffaut, Avignon
  - Hopital Nord Franche Comté, Belfort
  - CHU Besancon, Besançon
  - CH Germon et Gauthier, Beuvry
  - Hopital Avicenne, Bobigny
  - CHU Pellegrin, Bordeaux
  - Hopital St-Andre, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier fleyriat, Bourg-en-Bresse
  - HIA Clermont Tonnerre, Brest
  - CHRU de la Cavale Blanche, Brest
  - CHU Caen, Caen
  - Centre Hospitalier Jean Rougie, Cahors
  - CH Charleville, Charleville-Mézières
  - Hopital Antoine Beclere, Clamart
  - HIA Percy, Clamart
  - Hopital Louis Mourier, Colombes
  - Centre Hospitalier Compiègne Noyon, Compiègne
  - Groupe Hospitalier Sud Ile de France, Corbeil-Essonnes
  - CH Sud Francilien, Corbeil-Essonnes
  - Clinique des Cèdres, Cornebarrieu
  - CHU Henri Mondor, Créteil
  - Centre Hospitalier de Dax, Dax
  - Centre Hospitalier de Dieppe, Dieppe
  - CHU Dijon Bourgogne, Dijon
  - Centre Hospitalier de la Dracénie, Draguignan
  - Centre Hospitalier Victor Jousselin, Dreux
  - Hopital Simone Veil, Eaubonne
  - Centre Hospitalier Sud Essonne, Étampes
  - Centre Hospitalier Communal des Alpes du Sud, Gap
  - Hopital Raymond Poincare, Garches
  - Centre Hospitalier Avranche Granville, Granville
  - CHU Grenoble Alpes, Grenoble
  - Centre Hospitalier de Gueret, Guéret
  - Centre Hospitalier de Haguenau, Haguenau
  - Grand Hopital de l'Est Francilien, Jossigny
  - Centre Hospitalier des 2 Vallées, Juvisy-sur-Orge
  - CHU Réunion Saint Pierre, La Réunion
  - CHD Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier La Rochelle, La Rochelle
  - CH de Versailles, Le Chesnay
  - CHU Kremlin-Bicetre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - Hopital Roger Salengro, Lille
  - Centre hospitalier Saint Philibert, Lomme
  - Centre Hospitalier Bretagne Sud, Lorient
  - CH St-Joseph St-Luc, Lyon
  - HIA Desgenettes Lyon, Lyon
  - Groupe Hospitalier Edouard Herriot, Lyon
  - Hopital Francois Quesnay, Mantes-la-Jolie
  - Hopital Européen Marseille, Marseille
  - CHU Marseille Hopital Nord, Marseille
  - Hopital de la Timone, Marseille
  - CH de Meaux, Meaux
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - GHIRM, Montfermeil
  - CHU Lapeyronie, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Hopital Laennec, Nantes
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hopital l'Archet, Nice
  - CHU Nimes, Nîmes
  - CHR d'Orléans Hopital la Source, Orléans
  - Hopital St Louis, Paris
  - GH Diaconnesses Croix Saint Simon, Paris
  - La Pitié Salpetriere, Paris
  - Cochin, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Necker Enfants Malades, Paris
  - CHU Robert Debré, Paris
  - HEGP, Paris
  - Hopital Tenon, Paris
  - CH Francois Miterrand, Pau
  - CH Poissy, Poissy
  - CHU Poitiers, Poitiers
  - CH de Pontoise, Pontoise
  - CH de la Région d'Annecy, Pringy
  - CH Leon Binet, Provins
  - Hopital Privé Claude Galien, Quincy-sous-Sénart
  - CHRU Reims, Reims
  - CHG Rochefort, Rochefort
  - CH de St-Brieuc, Saint-Brieuc
  - Centre Cardiologique du Nord, Saint-Denis
  - Hopital Delafontaine, Saint-Denis
  - Clinique de l'Union, Saint-Jean
  - HIA Béjin, Saint-Mandé
  - Hopital Saint Clair, Sète
  - CH de St-Malo, St-Malo
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
  - CHRU Bretonneau, Tours
  - Hopital Privé du Vert Galan, Tremblay-en-France
  - Centre Hospitalier de Troyes, Troyes
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Hopital Jean Bernard, Valenciennes
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Centre hospitalier André Mignot, Versailles
  - Centre Hospitalier de Vichy, Vichy
  - Institut Gustave Roussy, Villejuif
  - HIA Robert Pique, Villenave-d'Ornon
  - Centre Hospitalier Lucie et Raymond Aubrac, Villeneuve-Saint-Georges
  - Hopital Privé du Val d'Yerres, Yerres

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] SRLF Trial Group. End of life in the critically ill patient: evaluation of experience of end of life by caregivers (EOLE study). Ann Intensive Care. 2021 Nov 26;11(1):162. doi: 10.1186/s13613-021-00944-z. PMID 34825996